CLINICAL TRIAL: NCT06875440
Title: A Comparison of Chlorhexidine and Green Tea Mouthwash in Patients With Gingivitis and Their Salivary Neutrophil and TAC Levels
Acronym: (1346)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Amirhossein Farahmand, Periodontist, Associate Professor, Department of Periodontics, Faculty of Dentistry, Tehran Medical Sciences, Islamic Azad University, Tehran, Iran, Affiliation: Islamic Azad University, Tehran, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1346
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Periodontal Diseases
Keywords: Gingivitis, Saliva, Green tea, Chlorhexidine, Neutrophil
MeSH Terms: conditions — Periodontal Diseases; Gingivitis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, Randomized, Double-blind, Controlled design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was carried out utilizing a double-blind approach. To guarantee objectivity, all three groups - the CHX group, the Green tea group, and the control group - received medications that were indistinguishable in terms of appearance, packaging, and color. Additionally, to minimize any potential bias, a clinician who had no association with the research labeled the medications as A and B, based on their content, and then distributed them among the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHX mouthwash (Experimental): Participants in Group A were administered CHX two times daily throughout the two-month study period. After the study concluded, the clinical periodontal parameters were reevaluated to assess any potential impact of the supplements on oral health.. To compare the total PMN level in saliva before and after the consumption of the Green tea mouthwash, as well as in individuals who did not receive any form of medication, 2 ml of non-stimulated saliva was collected from each participant at the commencement and conclusion of the study. These samples were then analyzed using UV-spectrophotometric methods to determine any variations in Neutrophil levels.
  Interventions: Drug: CHX mouthwash
- Green Tea mouthwash (Active Comparator): Participants in Group B were administered Green tea two times daily throughout the two-month study period. After the study concluded, the clinical periodontal parameters were reevaluated to assess any potential impact of the supplements on oral health.. To compare the total PMN level in saliva before and after the consumption of the CHX mouthwash, as well as in individuals who did not receive any form of medication, 2 ml of non-stimulated saliva was collected from each participant at the commencement and conclusion of the study. These samples were then analyzed using UV-spectrophotometric methods to determine any variations in Neutrophil levels.
  Interventions: Drug: CHX mouthwash

INTERVENTIONS:
Drug: CHX mouthwash — A total of 84 individuals diagnosed with gingivitis were selected for this study. These participants were randomly assigned to two different groups. The purpose of the study was to measure the periodontal parameters of the two molars adjacent to the mandible using a periodontal probe. All of the patients received scaling and root planing (SRP) as part of their treatment. However, the treatment groups differed in terms of the supplements they received. Group A was given a twice-daily dose of CHX, while Group B received a daily dose of Green tea. In addition to this, 2 ml of unstimulated saliva was collected from each patient both before and after 2 months. The purpose of collecting the saliva samples was to evaluate the total Neutrophil level and determine if there were any changes over time.
  Other Names: Green tea mouthwash

SUMMARY:
A Comparison of Chlorhexidine and Green Tea Mouthwash in Patients With Gingivitis and Their Salivary Neutrophil and TAC Levels.

DETAILED DESCRIPTION:
This research was structured as a double-blind, randomized clinical trial to assess the effectiveness of CHX and green tea mouthwash on periodontal health in patients with gingivitis. 84 patients from the Department of Periodontics at Broujerd Dental School of the Islamic Azad University of Medical Sciences were chosen for the study. Before the commencement of the trial, various clinical periodontal parameters, such as plaque index, bleeding on probing, gingival index, probing depth, and clinical attachment level, were measured in six different areas of the tooth surface. Subsequently, scaling and root planning were carried out, and oral hygiene practices were enhanced for all participants. The participants were then randomly divided into three groups: Group A, CHX, and Group B, which was provided with Green tea mouthwash two times daily. After three months, the clinical periodontal parameters were reevaluated. Furthermore, to compare the total PMN and TAC levels in saliva before and after the administration of these supplements, as well as in patients who did not receive any medication, 2 ml of non-stimulated saliva was collected from each participant at the beginning and end of the study for analysis using UV-spectrophotometric methods. The selection criteria for eligible participants in this study were also clearly defined.

ELIGIBILITY:
Inclusion Criteria:

a minimum of 20 natural teeth; a mean plaque index (PI) of at least 1.5, (10); a mean gingival index (GI) of at least 1.0 (Patients with a gingival index score of ≥1 at more than 60% of sites

Exclusion Criteria:

with systemic diseases, those who had undergone antibiotic therapy in the past three months, and anyone who had received periodontal treatment within the last six months. Participants diagnosed with aggressive periodontitis, individuals with known allergies to statin medications, and those currently undergoing statin treatment or using medications that may affect periodontal health were also not eligible. Furthermore, individuals who are immunocompromised, those who use tobacco products, and lactating or pregnant women were excluded from participation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-09-22 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Total Neutrophil level of saliva | 3 months
  UV-spectrophotometry was employed to assess the overall Neutrophil and TAC in saliva before and after consuming these supplements, as well as in individuals who were not administered any medication. A total of 2 ml of non-stimulated saliva was collected from each participant at the commencement and conclusion of the study for analysis using UV-spectrophotometric techniques.

SECONDARY OUTCOMES:
Plaque index | 3 months
  The evaluation of the plaque index will involve the utilization of a disclosing tablets, which will be used to compare the results with other groups at the beginning and end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Amirhossein Farahmand, Tehran, Tehran, Iran., Iran